CLINICAL TRIAL: NCT06782906
Title: Effect of Increased Physical Activity and Stopping Evening Snacking in Metabolic Health in Youth With Prediabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mustafa Tosur, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-56321; 58-3092-5-008 (Other Grant/Funding Number: USDA)
Record Dates: First submitted 2025-01-07; First posted 2025-01-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants in the intervention arm will be asked to perform ≥10,000 daily steps (≥5 days/week) and omit evening snacking after 8:00 p.m.
  Interventions: Behavioral: ≥10,000 daily steps (≥5 days/week) and stopping evening snacking
- Standard of Care Arm (No Intervention): Participants in the standard of care arm will be asked to follow recommendations of their physician.

INTERVENTIONS:
Behavioral: ≥10,000 daily steps (≥5 days/week) and stopping evening snacking — Participants in the intervention arm will be asked to perform ≥10,000 daily steps (≥5 days/week) and omit evening snacking after 8:00 p.m.
  Arms: Intervention Arm

SUMMARY:
Non-healthy eating habits and a lack of exercise contribute to prediabetes and type 2 diabetes (T2D). Evening snacking is linked to abnormal weight gain in adults and healthy adolescents. Most adolescents do not get enough exercise. This study aims to look at the benefits of more exercise and stopping evening snacking in youth with prediabetes. The study lasts 8 weeks, and participants will be randomly assigned to either an intervention group or a standard of care group.

DETAILED DESCRIPTION:
Poor nutrition in addition to a lack of physical activity play significant roles in childhood T2D development, primarily by negatively affecting adiposity and insulin action in concert with other T2D risk factors. Many aspects of nutrition, including frequency of eating, were examined in relation to obesity/increased adiposity and T2D risk. Previous studies suggest increased snacking may cause overeating, and potentially lead to weight gain.

Findings from adolescents in the 2005-2016 National Health and Nutrition Examination Survey (NHANES), showed those with overweight/obesity consume more snacks per day (1.85 and 1.97 snacks per day, respectively) and more calories per snack (305 and 340 kcal/snack, respectively) than their normal-weight peers (1.69 and 262 kcal/snack).Snack consumption in adolescents is also correlated with higher daily energy intake, lower fruit/vegetable intake, along with more frequent fast-food and sugar-sweetened beverage consumptions. The timing of snacking occasions has also emerged as a potential confounder. Among adults, greater evening snacking was associated with higher BMI and higher obesogenic dietary index (e.g., intake of fast food, etc.) while greater morning snacking was associated with increased fruit and vegetable consumption. Having a bedtime snack was associated with increased odds of overweight/obesity (1.47, 95% CI: 1.34-1.62) in Japanese women. Evening snacking was also shown to be independently correlated with overweight/obesity in Italian adolescents (RR 3.12, 95% CI: 1.17-8.34). In the Healthy Growth Study, children who had high-energy intake at dinner and evening snacking were more likely to skip breakfast - a metabolically unhealthy habit.

Also, despite the known metabolic benefits of physical activity, only 1 in 4 adolescents achieve recommended daily physical activity goals (60-min, moderate-to-vigorous physical activity (MVPA)/day).Both snacking and exercise may also affect metabolic health by independently modulating gene expression levels of critical metabolic pathways and subsequently intracellular signaling. Metabolic dysregulation resulting in altered plasma concentrations of several amino acids (e.g., higher branch-chain amino acid and lower glycine concentrations, etc.) was associated with insulin resistance.

Therefore, targeted interventions towards evening snacking and increased physical activity may prove beneficial in adolescents with prediabetes by preventing progression to T2D.

ELIGIBILITY:
Inclusion Criteria:

1. 12-18 years of age
2. Having a diagnosis of prediabetes
3. Engaging in frequent evening snacking
4. Inadequate physical activity

Exclusion Criteria:

1. Diagnosis of diabetes
2. Significant history of chronic disease
3. Evidence of significant liver or kidney disease;
4. Any hormone replacement therapy; and
5. Pregnancy.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity index for glucose disposal (ISI [Gly]) during oral glucose tolerance test | At week 9-10 following completion of 8 weeks of intervention period
  Insulin sensitivity index for glycemia (ISI [Gly]) will be calculated with a formula using insulin and glucose area under the curves during oral glucose tolerance tests (OGTT) as described previously (Belfiore et al., Metabolism, 2001):
  ISI (Gly) = 2 / [INSp x GLYp) + 1]
  INSp: insulinemic area during OGTT with 3 (0, 1h and 2h) or 5 sampling (0, 30, 60, 90 and 120 min) GLYp: glycemic area during OGTT (0, 1h and 2h) or 5 sampling (0, 30, 60, 90 and 120 min)
  INSp and GLYp are expressed by taking the mean normal value as 1, i.e., by dividing the value observed in the person under study by the mean normal value so that, if INSp (or GLYp) is 1.5-fold the mean normal values, it will be considered as equal to 1.5, and so on. We will use appropriate "mean normal values," which will be derived from data obtained in our laboratory.

SECONDARY OUTCOMES:
index for fat disposal (ISI [FFA]) during oral glucose tolerance test | At week 9-10 following completion of 8 weeks of intervention period
  Insulin sensitivity index for fat disposal (ISI [FFA]) will be calculated with a formula using insulin and free fatty acid area under the curves during oral glucose tolerance tests (OGTT) as described previously (Belfiore et al., Metabolism, 2001):
  ISI (FFA) = 2 / [INSp x FFAp) + 1]
  INSp: insulinemic area during OGTT with 3 (0, 1h and 2h) or 5 sampling (0, 30, 60, 90 and 120 min) FFAp: glycemic area during OGTT (0, 1h and 2h) or 5 sampling (0, 30, 60, 90 and 120 min)
  INSp and FFAp are expressed by taking the mean normal value as 1, i.e., by dividing the value observed in the person under study by the mean normal value so that, if INSp or FFAp) is 1.5-fold the mean normal values, it will be considered as equal to 1.5, and so on. We will use appropriate "mean normal values," which will be derived from data obtained in our laboratory.
HbA1c | At week 9-10 following completion of 8 weeks of intervention period
  Hemoglobin A1c (HbA1c) as measured in the plasma.
Percentage of adiposity (percent body fat) | At week 9-10 following completion of 8 weeks of intervention period
  Percent body fat as measured by DXA scan
Amino acid concentrations | At week 9-10 following completion of 8 weeks of intervention period
  Fasting amino acid concentrations as measured in the plasma
Adiponectin | At week 9-10 following completion of 8 weeks of intervention period
  Fasting adiponectin concentration as measured in the plasma
C-reactive protein (CRP) | At week 9-10 following completion of 8 weeks of intervention period
  CRP concentration as measured in the plasma
TNF-alpha | At week 9-10 following completion of 8 weeks of intervention period
  TNF-alpha concentrations as measured in the plasma
Interleukin 6 (IL-6) | At week 9-10 following completion of 8 weeks of intervention period
  IL-6 level as measured in the plasma
Gene expression levels of critical pathways | At week 9-10 following completion of 8 weeks of intervention period
  RNA sequencing for gene expression levels of critical metabolic pathways
Total energy expenditure | At week 9-10 following completion of 8 weeks of intervention period
  In a subset of cohort (n=20), free-living total energy expenditure (TEE) will be measured by the doubly labeled water (DLW) over a 14-d period using multiple urine collections at different time points. This optional part will be offered to all participants, and similar number of participants will be selected randomly from both arms (intervention and standard of care arm) by balancing gender and age categories.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Tosur, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital / Children's Nutrition Research Center / Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No